CLINICAL TRIAL: NCT00326716
Title: A Study of the Pharmacokinetics of Atazanavir (ATV)/Ritonavir(RTV) Administered as Part of Highly Active Antiretroviral Therapy (HAART) in HIV-1 Infected Pregnant Women
Brief Title: Pharmacokinetics of Atazanavir/Ritonavir in HIV-1 Infected Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-182
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: HIV Infection
Keywords: HIV-1 infected pregnant women, either treatment naive or on ATV/RTV combined with ZDV/3TC
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Atazanavir + Ritonavir + Combivir

INTERVENTIONS:
Drug: Atazanavir + Ritonavir + Combivir — Capsules, tablets, Oral, initially ATV 300 mg + RTV 100 mg + ZDV/3TC 300/150 mg, dose escalated to ATV 400 mg + RTV 100 mg + ZDV/3TC 300/150 mg, ATV and RTV once daily, lamivudine (ZDV) / zidovudine (3TC) twice daily (BID), up to 36 weeks
  Other Names: Reyataz; BMS-232632

SUMMARY:
To determine what dosing regimen of atazanavir (ATV) / ritonavir (RTV) produces adequate drug exposure during pregnancy compared to drug exposure in historical data in human immunodeficiency virus (HIV) infected participants.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected pregnant women
* > 18 years of age
* Between week 12 and 32 gestation
* CD4 > 200 cells/mm³
* Treatment-naive with HIV RNA > 400 c/mL, on HAART with HIV RNA <50 c/mL, or previously treated with ATV (< 3 weeks) with HIV RNA>400 c/mL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (2):
  - Triple O Medical Services, P.A., West Palm Beach, Florida
  - Women's Hospital Of Texas, Houston, Texas
- Local Institution, San Juan, Puerto Rico
- South Africa (3):
  - Local Institution, Soweto, Gauteng
  - Local Institution, Sunnyside, Gauteng
  - Local Institution, Westdene, Gauteng

REFERENCES:
- [Derived] Xu XS, Rose A, Demers R, Eley T, Ryan J, Stouffer B, Cojocaru L, Arnold M. Quantitative determination of free/bound atazanavir via high-throughput equilibrium dialysis and LC-MS/MS, and the application in ex vivo samples. Bioanalysis. 2014;6(23):3169-82. doi: 10.4155/bio.14.251. PMID 25529885
- [Derived] Eley T, Huang SP, Conradie F, Zorrilla CD, Josipovic D, Botes M, Osiyemi O, Hardy H, Bertz R, McGrath D. Clinical and pharmacogenetic factors affecting neonatal bilirubinemia following atazanavir treatment of mothers during pregnancy. AIDS Res Hum Retroviruses. 2013 Oct;29(10):1287-92. doi: 10.1089/AID.2013.0002. Epub 2013 Jul 19. PMID 23782005
- [Derived] Conradie F, Zorrilla C, Josipovic D, Botes M, Osiyemi O, Vandeloise E, Eley T, Child M, Bertz R, Hu W, Wirtz V, McGrath D. Safety and exposure of once-daily ritonavir-boosted atazanavir in HIV-infected pregnant women. HIV Med. 2011 Oct;12(9):570-9. doi: 10.1111/j.1468-1293.2011.00927.x. Epub 2011 May 16. PMID 21569187
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant participants were enrolled at 6 sites: United States (2), South Africa (3), and Puerto Rico (1).
Pre-assignment Details: Of the 69 enrolled participants, 28 mothers were not treated. Failure to continue to meet enrollment criteria resulting in discontinuation in 24/28 participants and 4 were not treated: 1 poor/no compliance, 1 met exclusion criteria, 1 was ARV naive subject with HIV RNA < 400 c/mL, and 1 was unable to comply with study procedures.
Groups:
- Mother ATV 300 mg / RTV 100 mg: Mothers receiving atazanavir (ATV) / ritonavir (RTV) 300/100 mg once daily (QD) + lamivudine (ZDV) / zidovudine (3TC) 300/150 mg twice daily (BID) during the third trimester. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Mother ATV 400 mg / RTV 100 mg: Mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID during the third trimester. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Infants ATV 300 mg / RTV 100 mg: Infants born to mothers receiving treatment with ATV 300 mg / RTV 100 mg during the third trimester of pregnancy.
- Infants ATV 400 mg / RTV 100 mg: Infants born to mothers receiving treatment with ATV 400 mg / RTV 100 mg during the third trimester of pregnancy.
Period: Pre-Natal Mothers
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg | Infants ATV 300 mg / RTV 100 mg | Infants ATV 400 mg / RTV 100 mg
Started | 20 | 21 | 0 | 0
Completed | 19 (Completion was defined as completing the study.) | 19 (Completion was defined as completing the study.) | 0 (Completion was defined as completing all follow up visits through 6 months.) | 0 (Completion was defined as completing all follow up visits through 6 months.)
Not Completed | 1 | 2 | 0 | 0
Not completed — Discontinued ATV Before Delivery | 1 | 2 | 0 | 0
Period: Infants
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg | Infants ATV 300 mg / RTV 100 mg | Infants ATV 400 mg / RTV 100 mg
Started | 0 | 0 | 20 (All infants were followed.) | 20 (All infants were followed. One mother withdrew consent pre-delivery and her infant was not followed.)
Completed | 0 | 0 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mother ATV 300 mg / RTV 100 mg: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during the third trimester. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Total: Total of all reporting groups
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age Continuous [Median (Full Range); unit: Years] | 29 [21 to 38] | 28 [19 to 37] | 28 [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 19 | 36
  White | 3 | 1 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 6 | 6 | 12
  Africa | 14 | 15 | 29
HIV RNA Distribution at Baseline [Number; unit: c/mL]
  <50 | 3 | 1 | 4
  50 to < 30,000 | 13 | 13 | 26
  30,000 to < 100,000 | 3 | 6 | 9
  >= 100,000 | 1 | 1 | 2
Infant Gestational Age at Delivery [Median (Full Range); unit: Weeks] | 38 [35 to 40] | 38 [35 to 41] | 38 [35 to 41]

OUTCOME MEASURES:

1. Secondary Outcome: Maternal HIV Ribonucleic Acid (RNA) Level on Day of Delivery
Description: The maternal HIV RNA level is assessed by the Roche Amplicor® Ultrasensitive Assay Version 1.5.
Time Frame: Day of Delivery ± 2 Days
Population: The analysis for the proportion of HIV RNA < 400 and < 50 c/mL at delivery is based on the Virologic Response - Observed Cases (VR-OC). VR-OC classifies subjects who remain on study therapy as responders according to a single HIV RNA measurement < 400 c/mL (or < 50 c/mL) closest to delivery and within delivery date ± 2 days.
Measure: Number; unit: Participants
Groups:
- Mothers ATV 300 mg / RTV 100 mg: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 38 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Mothers ATV 400 mg / RTV 100 mg: Mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 36 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / RTV 100 mg | Mothers ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 19 | 20
Participants
  HIV RNA < 400 copies/mL | 19 | 20
  HIV RNA < 50 copies/mL | 19 | 19

2. Secondary Outcome: Median Change From Baseline to Day of Delivery in Maternal HIV RNA Level
Description: The maternal HIV RNA level was determined at baseline and the day of delivery ± 2 days using VR-OC. The maternal HIV RNA level is assessed by the Roche Amplicor® Ultrasensitive Assay Version 1.5.
Time Frame: Baseline, Day of Delivery ± 2 Days
Population: The median maternal HIV RNA Level Change From Baseline was calculated for all treated mothers at the time of delivery. The maternal HIV RNA level at delivery was determined as the closest to delivery and within a pre-defined visit window for delivery, which is delivery date ± 2 days.
Measure: Median (Inter-Quartile Range); unit: log10 c / mL
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 18 | 19
log10 c / mL | -1.8 [-2.43 to -1.39] | -2.37 [-2.93 to -1.81]

3. Secondary Outcome: Mean HIV RNA Level at Baseline
Time Frame: Baseline
Population: All treated participants.
Measure: Mean (Standard Error); unit: log10 cm / mL
Groups:
- Mothers ATV 300 mg / RTV 100 mg Third Trimester: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 36 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Mothers ATV 400 mg / RTV 100 mg Third Trimester: Mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 36 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 20 | 21
log10 cm / mL | 3.520 (0.232) | 4.020 (0.171)

4. Secondary Outcome: Median Change From Baseline to Day of Delivery in Maternal Cluster of Differentiation 4 (CD4) Cell Count
Description: The median CD4 cell count change from baseline was calculated for all treated mothers at the time of delivery ± 2 days. Maternal CD4 cell counts were assessed by the Roche Amplicor® Ultrasensitive Assay Version 1.5.
Time Frame: Baseline, Day of Delivery ± 2 Days
Population: The median CD4 Cell Count Change From Baseline was calculated based on all treated mothers. The maternal CD4 cell count at delivery was determined as the closest to delivery and within a pre-defined visit window for delivery, which is delivery date ± 2 days.
Measure: Median (Inter-Quartile Range); unit: cells / mm^3
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 17 | 20
cells / mm^3 | 89 [-75 to 213] | 174 [-39 to 257]

5. Secondary Outcome: Mean CD4 Cell Count at Baseline
Time Frame: Baseline
Population: All treated participants.
Measure: Mean (Standard Error); unit: cells / mm^3
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 20 | 21
cells / mm^3 | 435.0 (39.2) | 390.0 (25.0)

6. Secondary Outcome: Infant HIV Status
Description: The neonatal HIV-1 status are assessed by the Roche Amplicor HIV-1 DNA Assay Version 1.5 (Roche Molecular Systems).
Time Frame: Birth Through 6 Months on Study
Population: All infants.
Measure: Number; unit: Participants
Arm/Group | Infant ATV 300 mg / RTV 100 mg | Infant ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 20
Participants
  HIV Positive | 0 | 0
  HIV Negative | 20 | 20

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE =any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: During study period and 30 days post-study.
Population: The number of SAEs is based on enrolled participants. Data were pooled from the ATV 300 mg / RTV 100 mg and ATV 400 mg / RTV 100 mg groups for all treated mothers and all infants.
Measure: Number; unit: Participants
Groups:
- All Treated Mothers: Data are pooled for mothers in the ATV 300 mg / RTV 100 mg and the ATV 400 mg / 100 mg groups.
- All Infants: Data are pooled for infants in the ATV 300 mg / RTV 100 mg and the ATV 400 mg / 100 mg groups.
Arm/Group | All Treated Mothers | All Infants
Number analyzed (Participants) | 41 | 40
Participants
  Death (n=41, n=40) | 0 | 0
  Serious Adverse Event (n=41, n=40) | 16 | 14
  Total AEs Leading to Discontinuation (n=41, n=40) | 2 | 2
  Anemia Leading to Discontinuation (n=41, n=40) | 1 | 2
  Transaminitis Discontinuation (n=41, n=40) | 1 | 0
  Prematurity Causing Discontinuation (n=41, n=40) | NA — Prematurity causing discontinuation was considered an infant only AE/SAE and thus was not deemed appropriate for evaluation in the mothers only population. | 1
  All AEs (n=41, n=40) | 40 | 40
  Anemia (n=41, n=40) | 6 | 3
  Diarrhea (n=41, n=40) | 4 | 4
  Nausea (n=41, n=40) | 6 | 0
  Vomiting (n=41, n=40) | 7 | 5
  Jaundice (n=41, n=40) | 10 | 20
  Hyperbilirubinemia (n=41, n=40) | 1 | 1
  Ocular Icterus (n=41, n=40) | 3 | 0
  Skin / subcutaneous tissue disorders (n=41, n=40) | 10 | 20

8. Secondary Outcome: Number of Participants With Grade 2 to Grade 4 AEs and SAEs
Description: AEs and SAEs considered possibly, probably, or certainly related to study treatment, were graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death). Hyperbilirubinemia (Grade 1=1.1 to 1.5 upper limit of normal [ULN] [mild], Grade 2=1.6 to 2.5 ULN [moderate], Grade 3=2.6 to 5.0 ULN [severe], Grade 4= > 5.0 ULN [potentially life threatening]).
Time Frame: During Study Period and 30 Days Post-Study.
Population: Data were pooled from the ATV 300 mg / RTV 100 mg and ATV 400 mg / RTV 100 mg groups for all treated mothers and all infants. The number of AEs and SAEs is based on enrolled participants.
Measure: Number; unit: Participants
Arm/Group | All Treated Mothers | All Infants
Number analyzed (Participants) | 41 | 40
Participants
  Grade 2 to Grade 4 (n=41, n=40) | 32 | 19
  Related Grade 2 to Grade 4 (n=41, n=40) | 10 | 0
  Grade 3 to Grade 4 (n=41, n=40) | 12 | 8
  Grade 3 to Grade 4 Total Bilirubin (n=41, n=40) | 19 | 7

9. Secondary Outcome: SAEs in Enrolled Mothers
Description: SAEs were evaluated for all treated and untreated participants. An SAE was defined as an untoward medical occurrence that results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event); might have caused death if it were more severe, required inpatient hospitalization or prolongation of existing hospitalization, in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, an important medical event that required intervention to prevent serious outcomes.
Time Frame: During Study Period and 30 Days Post-Study.
Population: Data were analyzed for all treated and untreated mothers.
Measure: Number; unit: Participants
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 21
Participants
  Any Adverse Experience | 7 | 8
  Blood and Lymphatic System Disorders | 1 | 2
  Anemia | 1 | 2
  Cardiac Disorders | 1 | 1
  Cardiomyopathy | 1 | 0
  Sinus Arrhythmia | 0 | 1
  Gastrointestinal Disorders | 0 | 1
  Abdominal Hernia | 0 | 1
  Hepatobiliary Disorders | 0 | 1
  Hyperbilirubinemia | 0 | 1
  Infections and Infestations | 2 | 2
  Endometrial Decidual | 2 | 0
  Pneumonia | 0 | 1
  Sepsis | 0 | 1
  Investigations | 0 | 1
  Transaminases Increased | 0 | 1
  Pregnancy, Puerperium, and Perinatal Conditions | 2 | 2
  Amenorrhea | 0 | 1
  Pre-eclampsia | 1 | 1
  Pregnancy Induced Hypertension | 0 | 0
  Premature Rupture of Membranes | 1 | 0
  Vascular Disorders | 1 | 1
  Hypertension | 0 | 1
  Hemorrhage | 1 | 0

10. Secondary Outcome: SAEs in Enrolled Infants
Description: as for outcome 9
Time Frame: Birth Through Week 16 of Life
Population: SAEs were recorded for all enrolled infants.
Measure: Number; unit: Participants
Groups:
- Infant ATV 300 mg / RTV 100 mg: Infants of mothers taking ATV 300 mg / RTV 100 mg at birth.
- Infant ATV 400 mg / RTV 100 mg: Infants of mothers taking ATV 400 mg / RTV 100 mg at birth.
Arm/Group | Infant ATV 300 mg / RTV 100 mg | Infant ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 20
Participants
  Any Adverse Experience | 10 | 4
  Blood and Lymphatic System Disorders | 1 | 1
  Anemia | 1 | 1
  Cardiac Disorders | 1 | 0
  Cardio-Respiratory Arrest | 1 | 0
  Restrictive Cardiomyopathy | 1 | 0
  Congenital, Familial, and Genetic Disorders | 0 | 1
  Atrial Septal Defect | 0 | 1
  Gastrointestinal Disorders | 1 | 0
  Constipation | 1 | 0
  Vomiting | 1 | 0
  Hepatobiliary Disorders | 1 | 1
  Hyperbilirubinemia | 0 | 1
  Jaundice | 1 | 0
  Infections and Infestations | 4 | 2
  Bronchiolitis | 0 | 2
  Gastroenteritis | 1 | 0
  Meningitis | 1 | 0
  Pneumonia | 0 | 1
  Sepsis | 1 | 0
  Syphilis | 1 | 0
  Injury, Poisoning, and Procedural Complications | 1 | 0
  Overdose | 1 | 0
  Metabolism and Nutrition Disorders | 1 | 1
  Hyperkalemia | 1 | 0
  Hypoglycemia | 0 | 1
  Nervous System Disorders | 1 | 0
  Cerebral Ischemia | 1 | 0
  Convulsion | 1 | 0
  Pregnancy, Puerperium, and Perinatal Conditions | 1 | 1
  Premature Baby | 1 | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 2 | 0
  Neonatal Respiratory Distress Syndrome | 1 | 0
  Respiratory Distress | 1 | 0

11. Primary Outcome: Infant Gestational Age at Delivery
Time Frame: At the time of delivery
Population: All infants.
Measure: Mean (Standard Error); unit: Weeks
Groups:
- Mothers ATV 300 mg / 100 mg Third Trimester: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 38 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Mothers ATV 400 mg / 100 mg Third Trimester: Mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 28 to 36 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 20 | 20
Weeks | 38 (0.3) | 38 (0.3)

12. Primary Outcome: Infant Gender
Time Frame: At the time of delivery
Population: All infants.
Measure: Number; unit: Participants
Arm/Group | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 20 | 20
Participants
  Male | 12 | 9
  Female | 8 | 11

13. Primary Outcome: Infant Race
Time Frame: At the time of delivery
Population: All infants.
Measure: Number; unit: Participants
Arm/Group | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 20 | 20
Participants
  Black | 15 | 18
  White | 5 | 1
  Mixed Race | 0 | 1

14. Primary Outcome: Mean ATV Maximum Plasma Concentration (Cmax) in One Dosing Interval
Description: Cmax = maximum observed plasma concentration of atazanavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the pharmacokinetic (PK) concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng / mL
Groups:
- Mothers ATV 300 mg / RTV 100 mg Second Trimester: Mothers receiving ATV/RTV 300/100 mg once daily (QD) + ZDV/3TC 300/150 mg twice daily (BID) during weeks 12 to 28 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng / mL | 3,729.09 [2,744.17 to 5,067.52] | 3,291.46 [2,444.82 to 4,431.30] | 4,210.76 [3,369.46 to 5,262.11]

15. Primary Outcome: Mean RTV Maximum Plasma Concentration (Cmax) in One Dosing Interval
Description: Cmax = maximum observed plasma concentration of ritonavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng / mL
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng / mL | 530.81 [333.20 to 845.61] | 587.36 [423.55 to 814.52] | 524.48 [368.76 to 745.95]

16. Primary Outcome: Mean ATV Area Under the Concentration Curve (AUC TAU)
Description: AUC = area under the concentration curve (AUC [TAU]) of atazanavir in one dosing interval from time zero to 24 hours.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng•h / mL
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng•h / mL | 34,399.13 [25,975.68 to 45,554.15] | 34,251.50 [27,173.69 to 43,172.84] | 46,602.45 [36,445.75 to 59,589.63]

17. Primary Outcome: Mean RTV Area Under the Concentration Curve (AUC TAU)
Description: AUC = area under the concentration curve (AUC [TAU]) of ritonavir in one dosing interval.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng•h / mL
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng•h / mL | 4,500.03 [3,243.97 to 6,242.43] | 4,664.93 [3,670.14 to 5,929.35] | 4,383.30 [3,107.41 to 6,183.06]

18. Primary Outcome: Mean ATV Trough Plasma Concentration (Cmin) 24 Hours Following the Daily Dose
Description: Cmin = plasma concentration 24 hours post dose of atazanavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum at 24 hours following the daily dose.
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng•h / mL
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng•h / mL | 663.78 [492.65 to 894.35] | 668.48 [529.06 to 844.64] | 916.63 [665.77 to 1,262.02]

19. Primary Outcome: Mean RTV Trough Plasma Concentration (Cmin) 24 Hours Following the Daily Dose
Description: Cmin = plasma concentration 24 hours post dose of ritonavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum at 24 hours following the daily dose.
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: ng•h / mL
Arm/Group | Mothers ATV 300 mg / RTV 100 mg Second Trimester | Mothers ATV 300 mg / RTV 100 mg Third Trimester | Mothers ATV 400 mg / RTV 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
ng•h / mL | 50.10 [28.39 to 88.43] | 41.12 [29.06 to 58.21] | 38.05 [26.24 to 55.17]

20. Primary Outcome: Mean ATV Terminal Elimination Half Life (T 1/2)
Description: T 1/2 = terminal elimination half life of atazanavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Groups:
- Mothers ATV 300 mg / 100 mg Second Trimester: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during weeks 12 to 28 of pregnancy. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / 100 mg Second Trimester | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
Hours | 10.42 [9.14 to 11.89] | 12.10 [9.44 to 15.51] | 12.17 [10.42 to 14.21]

21. Secondary Outcome: Mean Atazanavir Maternal Plasma Concentration and Neonatal Cord Blood Concentration
Description: Mean atazanavir maternal plasma concentration and neonatal cord blood concentration as measured at the time of delivery.
Time Frame: At Time of Delivery
Measure: Mean (Standard Deviation); unit: ng / mL
Groups:
- Mothers ATV 300 mg / RTV 100 mg: Mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID at the time of delivery. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Mothers ATV 400 mg / RTV 100 mg: Infants born to mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID at the time of delivery. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Mothers ATV 300 mg / RTV 100 mg | Mothers ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 21
ng / mL
  Maternal Serum Concentration | 1,412.05 (888.85) | 1,568.06 (846.44)
  Cord Blood Concentration | 273.20 (182.04) | 231.49 (158.29)

22. Secondary Outcome: Median Infant Total Bilirubin Level
Description: Median infant total bilirubin level as measured at specified time points.
Time Frame: Birth (Day 1), Day 3, Day 5, and Day 7 of Life
Measure: Median (Inter-Quartile Range); unit: mg / dL
Groups:
- Infant ATV 300 mg / RTV 100 mg: Infants of mothers receiving ATV/RTV 300/100 mg QD + ZDV/3TC 300/150 mg BID during the third trimester. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
- Infant ATV 400 mg / RTV 100 mg: Infansts of mothers receiving ATV/RTV 400/100 mg QD + ZDV/3TC 300/150 mg BID during the third trimester. Each dose of ATV/RTV (taken with a light meal or snack) was taken approximately 24 hours apart. Each dose of ZDV/3TC (taken with or without food) was taken approximately 12 hours apart.
Arm/Group | Infant ATV 300 mg / RTV 100 mg | Infant ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 20
mg / dL
  Day 1 (Birth) | 3.20 [2.80 to 4.30] | 3.25 [2.80 to 4.40]
  Day 3 | 8.40 [5.40 to 11.30] | 9.20 [7.00 to 9.60]
  Day 5 | 7.10 [3.05 to 10.20] | 9.25 [5.50 to 10.45]
  Day 7 | 5.10 [1.90 to 8.90] | 7.30 [2.50 to 9.30]

23. Secondary Outcome: Mean Atazanavir Plasma Protein Binding
Description: Atazanavir Plasma Protein Binding Percentage measured at specified time points.
Time Frame: Pregnancy Weeks 28 to Delivery at 3 Hours Postdose and 24 Hours Postdose, and Time of Delivery
Measure: Mean (Standard Deviation); unit: Percentage Bound
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 21
Percentage Bound
  Third Trimester 3 Hours Post Dose (n = 20, 20) | 91.34 (2.32) | 87.70 (2.69)
  Third Trimester 24 Hours Post Dose (n = 19, 20) | 90.37 (2.58) | 88.89 (2.40)
  Time of Delivery (n = 15, 12) | 77.05 (6.88) | 75.62 (4.34)

24. Secondary Outcome: Multicenter AIDS Cohort Study (MACS) Participant Adherence to Regimen and Drug Components for ATV 300 mg / RTV 100 mg Test Dose
Description: The MACS was administered to evaluate participant adherence to each drug and the adherence to the regimen. The MACS adherence questionnaire asks patients how many medication doses they missed during the previous day, 2 days, 3 days and 4 days. Drug-specific questions included adherence with dose and frequency. Adherence was defined as taking all doses and numbers of pills as prescribed for each medication. This strict adherence cut-off was based on the guidelines stating that anything less than excellent adherence may result in a virus breakthrough and development of resistance.
Time Frame: Study Week 2, Pregnancy Weeks 20 to Weeks 28, Pregnancy Weeks 28 to Delivery, Week 2 Postpartum, Week 4 Postpartum
Population: All treated participants were included in this evaluation.
Measure: Number; unit: Participants
Arm/Group | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Number analyzed (Participants) | 20 | 21
Participants
  Study Week 2 Regimen (n = 20,18) | 20 | 17
  Study Week 2 ATV (n = 20,18) | 20 | 17
  Study Week 2 RTV (n = 20,18) | 20 | 17
  Study Week 2 ZDV/3TC (n = 20,18) | 20 | 17
  Visit 1 Pregnancy Week 20 to 28 Regimen (n=12, 9) | 11 | 8
  Visit 1 Pregnancy Week 20 to 28 ATV (n=12, 9) | 12 | 8
  Visit 1 Pregnancy Week 20 to 28 RTV (n=12, 9) | 12 | 9
  Visit 1 Pregnancy Week 20 to 28 ZDV/3TC (n=12, 9) | 11 | 9
  Visit 2 Pregnancy Week 20 to 28 Regimen (n=8, 5) | 3 | 3
  Visit 2 Pregnancy Week 20 to 28 ATV (n=8, 5) | 8 | 5
  Visit 2 Pregnancy Week 20 to 28 RTV (n=8, 5) | 7 | 4
  Visit 2 Pregnancy Week 20 to 28 ZDV/3TC (n=8, 5) | 4 | 4
  Visit 3 Pregnancy Week 20 to 28 Regimen (n=6, 2) | 4 | 2
  Visit 3 Pregnancy Week 20 to 28 ATV (n=6, 2) | 5 | 2
  Visit 3 Pregnancy Week 20 to 28 RTV (n=6, 2) | 5 | 2
  Visit 3 Pregnancy Week 20 to 28 ADV/3TC (n=6, 2) | 4 | 2
  Visit 4 Pregnancy Wk 20 to 28 Regimen (n=0, 13) | NA — Participants were titrated to the ATV 400 mg / RTV 100 mg prior to this visit and thus data are not available for this dosing group. | 13
  Visit 4 Pregnancy Week 20 to 28 ATV (n=0, 13) | NA — Participants were titrated to the ATV 400 mg / RTV 100 mg prior to this visit and thus data are not available for this dosing group. | 13
  Visit 4 Pregnancy Week 20 to 28 RTV (n=0, 13) | NA — Participants were titrated to the ATV 400 mg / RTV 100 mg prior to this visit and thus data are not available for this dosing group. | 13
  Visit 4 Pregnancy Wk 20 to 28 ZDV/3TC (n=0, 13) | NA — Participants were titrated to the ATV 400 mg / RTV 100 mg prior to this visit and thus data are not available for this dosing group. | 13
  Visit 1 Pregnancy Wk 20 to Birth Regimen (n=20,20) | 19 | 20
  Visit 1 Pregnancy Week 20 to Birth ATV (n=20,20) | 20 | 20
  Visit 1 Pregnancy Week 20 to Birth RTV (n=20,20) | 20 | 20
  Visit 1 Pregnancy Wk 20 to Birth ZDV/3TC (n=20,20) | 19 | 20
  Visit 2 Pregnancy Wk 20 to Birth Regimen (n=19,19) | 18 | 18
  Visit 2 Pregnancy Week 20 to Birth ATV (n=19,19) | 19 | 19
  Visit 2 Pregnancy Week 20 to Birth RTV (n=19,19) | 19 | 19
  Visit 2 Pregnancy Wk 20 to Birth ZDV/3TC (n=19,19) | 18 | 18
  Visit 3 Pregnancy Wk 20 to Birth Regimen (n=15,19) | 12 | 18
  Visit 3 Pregnancy Week 20 to Birth ATV (n=15,19) | 13 | 19
  Visit 3 Pregnancy Week 20 to Birth RTV (n=15,19) | 13 | 19
  Visit 3 Pregnancy Wk 20 to Birth ZDV/3TC (n=15,19) | 12 | 18
  Visit 4 Pregnancy Wk 28 to Birth Regimen (n=5,15) | 5 | 15
  Visit 4 Pregnancy Week 28 to Birth ATV (n=5,15) | 5 | 15
  Visit 4 Pregnancy Week 28 to Birth RTV (n=5,15) | 5 | 15
  Visit 4 Pregnancy Wk 28 to Birth ZDV/3TC (n=5,15) | 5 | 15
  Visit 5 Pregnancy Wk 28 to Birth Regimen (n=1, 2) | 1 | 2
  Visit 5 Pregnancy Week 28 to Birth ATV (n=1, 2) | 1 | 2
  Visit 5 Pregnancy Week 28 to Birth RTV (n=1, 2) | 1 | 2
  Visit 5 Pregnancy Wk 28 to Birth ZDV/3TC (n=1, 2) | 1 | 2
  Visit 6 Pregnancy Wk 28 to Birth Regimen (n=0, 1) | NA — Participants experienced a dose escalation from ATV 300 mg / RTV 100 mg to ATV 400 mg / RTV 100 mg in the third trimester and thus this value was not calculated. | 1
  Visit 6 Pregnancy Week 28 to Birth ATV (n=0, 1) | NA — Participants experienced a dose escalation from ATV 300 mg / RTV 100 mg to ATV 400 mg / RTV 100 mg in the third trimester and thus this value was not calculated. | 1
  Visit 6 Pregnancy Week 28 to Birth RTV (n=0, 1) | NA — Participants experienced a dose escalation from ATV 300 mg / RTV 100 mg to ATV 400 mg / RTV 100 mg in the third trimester and thus this value was not calculated. | 1
  Visit 6 Pregnancy Wk 28 to Birth ZDV/3TC (n=0, 1) | NA — Participants experienced a dose escalation from ATV 300 mg / RTV 100 mg to ATV 400 mg / RTV 100 mg in the third trimester and thus this value was not calculated. | 1
  Postpartum Week 2 Regimen (n=19, 19) | 14 | 18
  Postpartum Week 2 ATV (n=18, 19) | 16 | 18
  Postpartum Week 2 RTV (n=18, 19) | 16 | 18
  Postpartum Week 2 ZDV/3TC (n =19, 19) | 14 | 18
  Postpartum Week 4 Regimen (n=17, 19) | 16 | 18
  Postpartum Week 4 ATV (n=17, 19) | 17 | 19
  Postpartum Week 4 RTV (n=17, 19) | 16 | 19
  Postpartum Week 4 ZDV/3TC (n=17, 19) | 17 | 18

25. Primary Outcome: Mean RTV Terminal Elimination Half Life (T 1/2)
Description: T 1/2 = terminal elimination half life of ritonavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Mothers ATV 300 mg / 100 mg Second Trimester | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
Hours | 5.03 [4.51 to 5.60] | 5.28 [4.73 to 5.90] | 5.10 [4.30 to 6.05]

26. Primary Outcome: Mean ATV Time of Maximum Observed Plasma Concentration (Tmax)
Description: Tmax = time to reach maximum observed plasma concentration of atazanavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Mothers ATV 300 mg / 100 mg Second Trimester | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
Hours | 3.68 [2.92 to 4.64] | 2.94 [2.36 to 3.65] | 3.30 [2.57 to 4.23]

27. Primary Outcome: Mean RTV Time of Maximum Observed Plasma Concentration (Tmax)
Description: Tmax = time to reach the maximum observed plasma concentration of ritonavir at specified time points.
Time Frame: Pregnancy Weeks 12 to 28, Weeks 28 to 36, and 4-6 Weeks Postpartum
Population: Treated participants in the PK concentration data set.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Mothers ATV 300 mg / 100 mg Second Trimester | Mothers ATV 300 mg / 100 mg Third Trimester | Mothers ATV 400 mg / 100 mg Third Trimester
Number analyzed (Participants) | 9 | 20 | 20
Hours | 6.11 [3.81 to 9.80] | 4.15 [3.12 to 5.54] | 4.63 [3.45 to 6.19]

ADVERSE EVENTS:
Arm/Group | Infant ATV 300 mg / RTV 100 mg | Infant ATV 400 mg / RTV 100 mg | Mother ATV 300 mg / RTV 100 mg | Mother ATV 400 mg / RTV 100 mg
Serious Adverse Events (participants affected / at risk) | 10/20 | 4/20 | 7/20 | 8/21
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20 | 20/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant ATV 300 mg / RTV 100 mg (N=20) | Infant ATV 400 mg / RTV 100 mg (N=20) | Mother ATV 300 mg / RTV 100 mg (N=20) | Mother ATV 400 mg / RTV 100 mg (N=21)
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 0 | 0
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0
HAEMORRHAGE (Vascular disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1 | 0 | 1
CONVULSION (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 1
SYPHILIS (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 1
MENINGITIS (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHIOLITIS (Infections and infestations) | 0 | 2 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0
ENDOMETRITIS DECIDUAL (Infections and infestations) | 0 | 0 | 2 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
AMNIORRHOEA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
NEONATAL RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infant ATV 300 mg / RTV 100 mg (N=20) | Infant ATV 400 mg / RTV 100 mg (N=20) | Mother ATV 300 mg / RTV 100 mg (N=20) | Mother ATV 400 mg / RTV 100 mg (N=21)
CONJUNCTIVITIS (Eye disorders) | 3 | 1 | 0 | 0
OCULAR ICTERUS (Eye disorders) | 0 | 0 | 2 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 1 | 0 | 0
CARDIAC MURMUR (Investigations) | 0 | 2 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1 | 0
CULTURE URINE POSITIVE (Investigations) | 0 | 0 | 1 | 0
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0 | 0 | 2 | 0
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 3 | 3
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 9 | 10 | 4 | 6
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 2 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 7 | 2
SCIATICA (Nervous system disorders) | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 3 | 1
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 4 | 2
VOMITING (Gastrointestinal disorders) | 1 | 3 | 5 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 3 | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 3 | 2
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 3 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2 | 2 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 | 3 | 0 | 0
TONGUE GEOGRAPHIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 2 | 0
PAROTID GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 4 | 1 | 0
IMPETIGO (Infections and infestations) | 1 | 0 | 0 | 0
MASTITIS (Infections and infestations) | 0 | 0 | 1 | 0
RHINITIS (Infections and infestations) | 0 | 3 | 0 | 2
INFLUENZA (Infections and infestations) | 0 | 1 | 1 | 2
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
BODY TINEA (Infections and infestations) | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 3
TRACHEITIS (Infections and infestations) | 0 | 0 | 1 | 0
CANDIDIASIS (Infections and infestations) | 1 | 2 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 2
ENDOMETRITIS (Infections and infestations) | 0 | 0 | 1 | 0
OTITIS MEDIA (Infections and infestations) | 3 | 1 | 0 | 1
SKIN CANDIDA (Infections and infestations) | 0 | 1 | 0 | 0
WOUND SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
BRONCHIOLITIS (Infections and infestations) | 2 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 1 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 2 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 3 | 3 | 2 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 2
VAGINITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 6
SKIN BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 10 | 8 | 4
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
GESTATIONAL DIABETES (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
HEAT RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
NAIL PIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 2 | 2
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
CONGENITAL NAEVUS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 1
PROLONGED LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
CAPUT SUCCEDANEUM (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
JAUNDICE NEONATAL (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
NEONATAL DISORDER (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
PREGNANCY INDUCED HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
JOINT HYPEREXTENSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
MASS (General disorders) | 0 | 1 | 0 | 0
PAIN (General disorders) | 0 | 0 | 1 | 1
FATIGUE (General disorders) | 0 | 0 | 4 | 0
PYREXIA (General disorders) | 1 | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.